CLINICAL TRIAL: NCT02682004
Title: Serotonin, Leptin and Adiponectin Level in Patients With Postpartum Depression: Controlled Study
Status: Completed | Type: Observational
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Baki Senturk, Principal investigator, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Other Study IDs: 51
Record Dates: First submitted 2016-02-10; First posted 2016-02-15 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Leptin; Serotonin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Women with postpartum depression
  Interventions: Other: leptin, serotonin and adiponectin level
- Women without postpartum depression
  Interventions: Other: leptin,serotonin, adiponectin level

INTERVENTIONS:
Other: leptin, serotonin and adiponectin level
  Groups: Women with postpartum depression
Other: leptin,serotonin, adiponectin level
  Groups: Women without postpartum depression

SUMMARY:
After vaginal delivery, all of the participants will evaluate by using Edinburg depression scale and venous blood sample will obtain. Postpartum depression will consider the result of scale 13 and above according to Turkhish translate. Then leptin, adiponectin and serotonin level will compare between depressed and nondepressed women.

ELIGIBILITY:
Inclusion Criteria:

* All women who gave birth

Exclusion Criteria:

* women with previously diagnosed depression and any psychiatric disorders
* women with previously take antidepressan and antipshycothic
* women giving birth to children with anomalies
* women with undertake surgery for peripartum hemorrhage

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: According to Edinburg depression scale womenn who taken 13 point and above.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-02; Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Blood level (ng/ml) ELİSA | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Maternity and Pediatric Research and Training Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Hu Y, Dong X, Chen J. Adiponectin and depression: A meta-analysis. Biomed Rep. 2015 Jan;3(1):38-42. doi: 10.3892/br.2014.372. Epub 2014 Oct 16. PMID 25469244
- [Result] Skalkidou A, Sylven SM, Papadopoulos FC, Olovsson M, Larsson A, Sundstrom-Poromaa I. Risk of postpartum depression in association with serum leptin and interleukin-6 levels at delivery: a nested case-control study within the UPPSAT cohort. Psychoneuroendocrinology. 2009 Oct;34(9):1329-37. doi: 10.1016/j.psyneuen.2009.04.003. Epub 2009 May 7. PMID 19427131
- [Result] Mansur RB, Rizzo LB, Santos CM, Asevedo E, Cunha GR, Noto MN, Pedrini M, Zeni M, Cordeiro Q, McIntyre RS, Brietzke E. Adipokines, metabolic dysfunction and illness course in bipolar disorder. J Psychiatr Res. 2016 Mar;74:63-9. doi: 10.1016/j.jpsychires.2015.12.003. Epub 2015 Dec 12. PMID 26748249
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/25469244
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=risk+of+postpartum+depression+in+association+with+serum+leptin+and
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/26748249